CLINICAL TRIAL: NCT01632709
Title: Pathophysiology of Post Amputation Pain
Acronym: PPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northwestern University (Other)
Responsible Party: Principal Investigator, Dr. Norman Harden, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOD_PAP 12
Record Dates: First submitted 2012-06-11; First posted 2012-07-03 (Estimated); Results first posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Amputation Stumps; Neuroma
MeSH Terms: conditions — Neuroma | interventions — Bupivacaine; Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sympathetic nerve block of bupivacaine (Active Comparator): Sympathetic nerve block of bupivacaine
  Interventions: Drug: Bupivacaine
- Dry needling at the sympathetic ganglion (Placebo Comparator): Placebo/ Dry needling at the sympathetic ganglion
  Interventions: Drug: Placebo
- Neuroma injection of bupivacaine (Active Comparator): Neuroma injection of bupivacaine
  Interventions: Drug: Bupivacaine
- dry needling at the neuroma (Placebo Comparator): Placebo/ dry needling at the neuroma
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine — one injection of 10ml of .25%
  Arms: Neuroma injection of bupivacaine; Sympathetic nerve block of bupivacaine
Drug: Placebo — Dry needling
  Other Names: Dry needling
  Arms: Dry needling at the sympathetic ganglion; dry needling at the neuroma

SUMMARY:
The purpose of this study is to see how Post Amputation Pain (PAP) affects the body and brain by using sensory testing (such as pinprick testing), taking pictures of your brain (using a functional magnetic resonance imaging (fMRI) machine) and biomedical interventions (such as an injection of pain medicine). All medicines and the fMRI machine used during this study are FDA approved. The investigators hope that by learning the causes of PAP, the investigators can help future amputees.

DETAILED DESCRIPTION:
Your participation in this study will last for 5 weeks and you will be asked to come to a total of 3 visits. The first visit will be during the first week of the study, the second visit during the second week of the study and the third (final) visit will be during the fifth (and final) week of the study. For your first visit you will have a physical examination with some sensory stimulation tests (such as vibration and pinprick tests), some questionnaires about your health and pain history, hot and cold sensory tests, and we will take thermal pictures of your body before and after receiving a quick electrical stimulus. You will also be trained on how to use the finger-span device to rate your pain during the second visit, and how to use an electronic pain diary to record your pain scores three times a day during the five weeks of the study.

The second visit will begin with questionnaires from the first visit and thermal images with a quick electrical stimulus. You will then be brought to an fMRI scanner room at Northwestern University. For an hour and fifteen minutes we will take pictures of your brain and these pictures will help us understand the changes in your brain relating to pain. You will then be put into one of four treatment groups randomly.

The study treatment that you will get will be decided randomly or by chance, like flipping a coin. Injections in this study will use the local anesthetic bupivacaine (a long lasting drug like the numbing agent novocaine used by dentists). This drug causes numbness, blocks pain and other nerve function near the injection site for 6-8 hours. Group 1 will get a sympathetic nerve block of bupivacaine, which changes how your nerves transmit pain, in either the neck or lower back (depending on where the amputation is located), Group 2 will get a placebo injection (no active medicine) in either the neck or lower back (depending on where the amputation is located), Group 3 will get a neuroma injection of bupivacaine (a neuroma is a group of nerves at the end of your residual limb), and Group 4 will get a placebo injection (no active medicine) at the neuroma. Some people get the bupivacaine injection and some people get the placebo injection so that we can compare the groups and see if the bupivacaine brings more, less or the same pain relief as a placebo injection. We scan your brain before the injection so that we can see how your brain responds to pain. We also scan your brain after the injection so that we can see if your brain responds differently to pain after the injection has been done.

You will know the location of your injection before you receive the treatment (neck, lower back or neuroma on your affected limb), but you will not know if you are getting a pain medication injection or placebo injection. Only the study doctors will know this information, and it can be told to you in case of an emergency. After the injection, you will have a second hour of brain scanning. After the scanning, you will be asked to complete some questionnaires, sensory tests, hot and cold temperature testing and we will take thermal pictures of your body before and after a quick electrical stimulus.

Your third visit will be four weeks after your second visit. For your third visit you will have the same questionnaires as during the first and second visits, sensory tests, hot and cold temperature testing and we will take thermal pictures of your body before and after a quick electrical stimulus.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Able to read and speak English and provide informed consent
3. Single Amputation, upper or lower.
4. Subject has chronic post amputation pain lasting longer than three months
5. Subject has healed amputation wounds
6. Pain must be ≥3 on a scale of 0-10, 0 being no pain, 10 being the worse pain imaginable.
7. If subjects pain is non-existent during fMRI scans, the subject needs to be willing to have their pain induced by targeting pain trigger points (for example, study's postdoctoral fellow would massage certain regions of the affected limb to trigger PAP).
8. Subject agrees to 1) Stop taking all aspirin seven days prior to their second visit (Bayer,Ecotrin,Alka Seltzer, etc.) 2) All inflammatory medications 48 hours prior to their second visit (Advil, Motrin, Indocin, Lodine , Ibuprofen, Aleve, Naproxen, etc. 3) Supplements such as Vitamin E and Fish Oil 48 hours prior to their second visit.
9. Subject agrees to continue other prescribed medications.
10. Subject is willing to have hypodermic needle injections and images taken of them (digital, thermal, and fMRI).
11. Able to understand and comply with all data collection methodology including electronic diary.
12. If female, is not pregnant and not currently attempting to conceive; if of childbearing potential, use of a highly effective method of birth control (as determined by Pl).

Exclusion Criteria:

1. Subject is allergic to Isovue 300 or amide-type local anesthetics such as bupivicaine, lidocaine, or mepivacaine.
2. Subject has a diagnosis of bleeding diathesis or an immune compromise.
3. Subject has pain that is more severe than their post amputation pain.
4. Subject has a clinical diagnosis of fibromyalgia.
5. Subject has metal shavings and or is frequently in an environment where there is metal work being done or significant amounts of metal shavings.
6. Subject has ferrous metal implants, aneurism clips, bioelectric devices, and other implants which can be affected by the magnetic field of the MRI.
7. Subject is claustrophobic.
8. Subject weighs more than 300 pounds.
9. Subject plans to start new pain treatments or therapies during the study (e.g. new pain medication, injections, PT, surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Harden, M.D., Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were not assigned to an arm until Visit 2 (randomization).
Period: Overall Study
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling at Sympathetic Ganglion | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Started | 4 | 3 | 5 | 4
Completed Visit 2 (Received Injection) | 4 | 2 | 5 | 3
Completed | 2 | 2 | 5 | 3
Not Completed | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling at Sympathetic Ganglion | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma | Total
Number analyzed (Participants) | 4 | 2 | 5 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (11.9) | 55 (8.5) | 50.4 (9.4) | 43.3 (7) | 53.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 3 | 5
  Male | 4 | 1 | 4 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 2 | 0 | 2 | 1 | 5
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Pain rating before and after injection on a 0-10 NRS pain scale (0=no pain, 10= worst pain imaginable)
Time Frame: Pain rating before and at 15 minutes and 1 hour post injection
Population: all available data was analyzed (some subjects did not complete all outcomes)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dry Needling; Dry Needling at the Neuroma: Placebo: Dry needling
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Number analyzed (Participants) | 3 | 2 | 5 | 3
units on a scale
  NRS-Phantom Limb Pain (15 minutes post) | -0.3 (2.3) | -2 (0) | -1 (2.3) | 1.3 (0.6)
  NRS-Phantom Limb Pain (1 hour post) | -3.5 (0.7) | -1 (1.4) | -0.3 (0.6) | 0 (0)
  NRS-Residual Limb Pain (15 minutes post) | -1.7 (1.5) | -1 (1.4) | -2.2 (3.5) | 0.7 (0.6)
  NRS-Residual Limb Pain (1 hour post) | -2 (2.8) | -0.5 (0.7) | 0.3 (1.5) | 3 (4.2)

2. Secondary Outcome: Change in Perceived Disability (PDI)
Description: The PDI is a seven-item validated instrument that assesses perceived disability in 7 key life areas. The Pain Disability Scale is a scale from 0-70 where 0= no disability and 70=the most disability
Time Frame: PDI collected pre injection and 1 week post injection
Population: all available data was analyzed (some subjects did not complete all outcomes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Number analyzed (Participants) | 2 | 2 | 5 | 3
units on a scale | -16.5 (10.6) | -21.5 (24.7) | -5.2 (12.7) | 13.0 (18.2)

3. Secondary Outcome: Change in Perceived Anxiety (PASS)
Description: The Pain Anxitey Symptoms Scale (PASS) is a validated instrument that assesses anxiety in.The PASS is a scale from 0-100 where 0= no anxiety and 100=the most anxiety
Time Frame: PASS collected pre injection and 1 week post injection
Population: all available data was analyzed (some subjects did not complete all outcomes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Number analyzed (Participants) | 2 | 2 | 5 | 3
units on a scale | -3.0 (8.5) | -36.5 (5.0) | -1.0 (17.4) | 11.3 (14.6)

4. Secondary Outcome: Change in Depression (CES-D 10)
Description: The Center for Epidemiologic Studies Short Depression Scale (CES-D 10) is a validated instrument that assesses depression. The CES-D 10 is a scale from 0-30 where 0= no depression and 30=the most depression
Time Frame: CES-D 10 collected pre injection and 1 week post injection
Population: all available data was analyzed (some subjects did not complete all outcomes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Number analyzed (Participants) | 2 | 2 | 5 | 3
units on a scale | -2.0 (2.8) | -4.0 (2.8) | -2.0 (6.5) | 3.3 (5.8)

5. Secondary Outcome: Pain Visual Analogue Scale (VAS)
Description: The Pain Visual Analogue Scale (VAS) is a scale from 0-100 where 0= no pain and 100=the worst pain
Time Frame: VAS collected pre injection and 1 week post injection
Population: all available data was analyzed (some subjects did not complete all outcomes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sympathetic Nerve Block of Bupivacaine | Dry Needling | Neuroma Injection of Bupivacaine | Dry Needling at the Neuroma
Number analyzed (Participants) | 2 | 2 | 5 | 3
units on a scale
  Change in VAS- Phantom Limb Pain | -8.5 (36.1) | -8.0 (8.5) | -4.4 (42.6) | 10.8 (14.8)
  Change in VAS-Residual Limb Pain | 3.0 (18.4) | -10.8 (7.4) | -9.5 (20.6) | 5 (22.6)

ADVERSE EVENTS:
Arm/Group | Placebo/Sham Injection | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No